CLINICAL TRIAL: NCT01236833
Title: Enteral Administration of Lactated Ringer's Solution in Neonates With Feeding Intolerance, a Randomized Controlled Trial
Brief Title: Lactated Ringer's Solution in Neonates With Feeding Intolerance
Acronym: LR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Louis Beaumier, The Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-225-PED
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Intestinal Disease; Feeding Disorder Neonatal
Keywords: Lactated Ringer's Solution; Isotonic Solution; Intestinal Disease; Feeding Intolerance; Necrotizing Enterocolitis; Newborn; Premature Infant
MeSH Terms: conditions — Intestinal Diseases; Enterocolitis, Necrotizing; Premature Birth | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fasting (No Intervention)
- Lactated Ringer's Solution (Active Comparator)
  Interventions: Drug: Lactated Ringer's Solution

INTERVENTIONS:
Drug: Lactated Ringer's Solution — 2.5 ml per kg every 3 hours, via nasogastric tube, orogastric tube or orally, until the infant reaches 80 ml/kg/day of milk feeding or for a maximum of 14 days
  Other Names: Lactated Ringer's
  Arms: Lactated Ringer's Solution

SUMMARY:
The objective of this study is determining if enteral administration of Lactated Ringer's solution (LR) in preterm infants with feeding intolerance enables for faster advancement of milk feeding than fasting.

DETAILED DESCRIPTION:
Feeding intolerance is a common problem in premature infants in the Neonatal Intensive Care Unit. Definition is clinical and based on abdominal distension, abdominal tenderness, emesis, change in gastric residuals, presence of blood in stool, and apnea with bradycardia.

Feeding intolerance is associated with serious complications: necrotizing enterocolitis, longer hospitalization and prolonged intravenous nutrition complications (e.g. sepsis, liver damage). Therefore, the investigators aim to achieve adequate enteral nutrition as soon as possible.

Because LR is a an amniotic fluid-like solution, it may improve gastro-intestinal function and avoid fasting, as well as its multiple problems (e.g. intestinal atrophy and decreased intestinal motility). LR was chosen as the test solution because of experience documenting its safe use in comparable groups: in newborn resuscitation parenterally, in amnioinfusion, and in bowel irrigation. Moreover, LR is similar in electrolytes composition to the experimental solution used in previous studies by Barney et al in neonates.

ELIGIBILITY:
Inclusion Criteria:

* Birth gestational age (GA) between 25 and 32 weeks
* Corrected gestational age less than 34 weeks
* Enteral feeding tolerated at a minimum of 10 ml/kg/day for a minimum of 48 hours
* Severe feeding intolerance, defined as a minimum of one or more of the following signs leading to withholding of milk feedings on two evaluations over 12 to 24 hours:

  1. Significant increased abdominal girth, as evaluated by the treatment team, with abdominal tenderness
  2. Visible enlarged bowel loops with abdominal tenderness
  3. Recurrent emesis leading to withhold feeds
  4. Gastric residuals in excess of one feeding, recurrent or with growing abdominal girth
  5. Visible blood in stools without anal etiology
* Documented informed consent for participation in the study

Exclusion Criteria:

* Infants who already reached full enteral feeds for 72 hours, in fact a minimum of 130 ml/kg/day enteral feeds without parenteral supplementation.
* Small for gestational age (SGA) (weight at or less than the 3rd percentile on the Fenton growth chart)
* NEC (Bell's stage II or higher, radiologic evidence of NEC, pneumatosis intestinalis or free intraperitoneal air)or history of NEC
* Gastric or intestinal occlusion (no transit, absent bowel sounds, incessant vomiting, bile stained vomiting or air fluid levels)
* Major congenital malformation
* Septic infants requiring therapeutic antibiotics or antimycotics (infants only on prophylactic antibiotics or antimycotics should not be excluded).
* Patients judged as being too ill to enroll in this study, as defined by a requirement for mechanical ventilation with >50% FIO2
* Patent Ductus Arteriosus requiring ibuprofen, indomethacin or ligature, until one week after the end of treatment
* Intraventricular Haemorrhage grade 3 or 4
* Hypernatremia ≥ 150 mmol/L

Min Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Average of the daily enteral caloric intake (in calories/kg/day) received over the 14 days after study entry | 14 days
  To measure enteral caloric intake, the volume of milk feeding, for each patient will be recorded daily and for 14 days. Unfortified milk and fortified milk are calculated as containing respectively 0.67 Cal/ml and 0.81 Cal/ml.

SECONDARY OUTCOMES:
Number of days to reach 130 ml/kg milk feeding | variable
Number of days to discontinue IV access | variable
Growth (weight, height, head circumference), increase % after 14 days and between study entry and discharge home | variable
Length of hospitalization | variable
Necrotizing enterocolitis | during the 14 day-study period and hospitalization
Electrolytes, bilirubin, serum urea nitrogen, creatinine and liver enzymes | 14 days
Infections | until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Gaelle Sadani, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Louis Beaumier, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - McGill University Health Center, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Background] Barney CK, Lambert DK, Alder SC, Scoffield SH, Schmutz N, Christensen RD. Treating feeding intolerance with an enteral solution patterned after human amniotic fluid: a randomized, controlled, masked trial. J Perinatol. 2007 Jan;27(1):28-31. doi: 10.1038/sj.jp.7211609. PMID 17180128